CLINICAL TRIAL: NCT04980352
Title: Multi-dimensional Signatures for Precisely Predicting the Response and Prognosis of Lung Cancer Patients
Acronym: Pred-lung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Wuhan TongJi Hospital (Other); Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1-12 V1.1
Record Dates: First submitted 2021-07-11; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Response; Prognosis
Keywords: Multi-dimensional Signatures; NGS; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: real world treatment by doctors — real world treatment by doctors

SUMMARY:
This study aims to determine the clinical effectiveness of multi-dimensional signatures in predicting response and prognosis of lung cancer patients. The study is a multi-center perspective research of treatment planning for patients with lung cancer. To characterize clinical effectiveness, the progression-free survival (PFS) and overall survival (OS) impacts of multi-dimensional signatures will be estimated.

DETAILED DESCRIPTION:
Multi-dimensional signatures, including NGS-based genotyping, and other essential detections such as immunohistochemistry (IHC), provides an opportunity to improve outcomes for patients by tailoring treatments to each individual's genomic profile. This is a multi-center single arm research study integrating multi-dimensional signatures into clinical decision-making for patients with lung cancer. The clinical effectiveness of multi-dimensional signatures is unknown in the real-world of clinics. To identify a counterfactual for Pred-lung approach, matching methods combined with administrative healthcare data will be used. The survival impacts of Pred-lung approach compared to usual care in matched controls will then be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally-advanced or metastasis lung cancer
* Life expectancy > 3 months

Exclusion Criteria:

* Age at diagnosis <18
* refuse to enroll

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally-advanced or metastasis lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 6 months
  Progression-free survival

SECONDARY OUTCOMES:
OS | through study completion, an average of 1 year
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) are available upon reasonable requests.